CLINICAL TRIAL: NCT03696017
Title: Opioid/Benzodiazepine Polydrug Abuse: Integrating Research on Mechanisms, Treatment and Policies
Brief Title: Opioid/Benzodiazepine Polydrug Abuse
Status: Recruiting | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor, Wayne State University
Other Study IDs: Polydrug Aim 2
Record Dates: First submitted 2018-09-26; First posted 2018-10-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Polysubstance Abuse
Keywords: Opioid Abuse; Benzodiazepine abuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients either newly admitted to Substance Use Disorder treatment in Wayne County, or in treatment longer but are using opioids (40 patients per group).
  Interventions: Other: Multi-domain assessment battery
- Group 2: Patients either newly admitted to Substance Use Disorder treatment in Wayne County, or in treatment longer but are using benzodiazepines (BZD) (40 patients per group).
  Interventions: Other: Multi-domain assessment battery
- Group 3: Patients either newly admitted to Substance Use Disorder treatment in Wayne County, or in treatment longer but are using BZD/opioid (40 patients per group).
  Interventions: Other: Multi-domain assessment battery

INTERVENTIONS:
Other: Multi-domain assessment battery — Assessments of emotion regulation, neurocognitive performance, pain, sleep, and substance use. There is no therapeutic intervention; all participants are already independently in treatment for their substance use disorder and we are simply assessing them at baseline visit and 3-month follow-up.

SUMMARY:
Benzodiazepine (BZD)/opioid polysubstance abuse (PSA) dramatically increases risks of overdose, disability and death; however, little is known about phenotypes that could be targeted to decrease this use and these associated risks.

The opioid abuse epidemic is generating unprecedented numbers of overdoses (OD) and deaths from prescribed and illegal sources (e.g. fentanyl combined with, or sold as, heroin). Yet, medical and epidemiological data suggest these adverse outcomes are not solely due to over-consumption of opioids.The FDA recognizes the health danger of BZD/opioid PSA, and issued labeling changes for prescribing BZDs and opioids. Impact of these changes is unclear and could be minimal if people obtain these substances illegally.

BZD abuse can be harmful alone or combined with opioids, as BZDs: (a) contribute to OD/death e.g. 31% of opioid OD-related deaths from 1999 to 2011 were related to coincident BZD use, BZD co-use is dose-dependently related to mortality and rates of BZD OD deaths have sharply increased. (b) exacerbate progression and adverse outcomes of opioid abuse. and (c) worsen behavioral impairment from opioids, increase rates of falls and fractures, motor vehicle accidents, and sleep-disordered breathing.

There has been limited systematic research of BZD/opioid PSA. This is a major gap because BZD are often co-prescribed with opioids (in 33 to 50% of cases) and are easily obtained illegally.

In response to these problems, there is an urgent need to obtain population-level, clinical pharmacology, and mechanistic data to test our unified hypothesis of dual-deficit in affective/hedonic regulation.

DETAILED DESCRIPTION:
Up to 120 patients who are currently in Substance Use Disorder treatment in Wayne County who use opioids, benzodiazepines (BZD), or both, will be assessed. Patients will be referred from the treatment regulator and local providers, and by advertisements in the community.

Participants will take part in one 6 hour face-to-face assessment during which they will undergo comprehensive assessments of both clinical (substance use, mental health) and hypothesis-driven measures (affective, neurocognitive, behavioral).

Participants must provide a supervised alcohol-free breath sample and a urine sample that will be screened for opioids, methadone, cocaine metabolites, BZDs, barbiturates, amphetamines.

Psychopathology: The Semi-Structured Clinical Interview for DSM-5 will be used to evaluate lifetime and current psychiatric and substance use disorders.

Affective dysregulation (inability to regulate emotions), neurocognition, pain and prescription misuse, insomnia, sleepiness, vigilance, and substance use will be assessed through the use of computerized measurements as well as paper and pencil questionnaires and face-to-face interviews.

Sample Size: Up to 120 total participant will be evaluated. This will offer greater statistical power to detect affective and neurocognitive effects than prior studies, including analysis of sex differences and correction for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Recently admitted and/or not clinically stable in treatment for Substance Use Disorder (SUD) in Wayne County
* Using opioids, benzodiazepines (BZD), or BZD/opioid.

Exclusion Criteria:

* Participants with current psychosis, bipolar disorder, or severe depression (i.e. severe psychiatric disorder)
* Individuals with serious neurological disorders, e.g. brain tumor, history of stroke, history of traumatic brain injury w/ loss of consciousness
* Cognitive impairment (IQ<80)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will either be newly admitted to Substance Use Disorder treatment, or in treatment longer but still occasionally using substances.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Psychopathology | Administered once during the baseline clinical assessment.
  Semi-Structured Clinical Interview for DSM (Face-to-face interview) Evaluates lifetime and current psychiatric and substance use disorders.
Beck Depression Inventory-II | Administered during the baseline clinical assessment, and at the 3-month follow-up visit.
  Questionnaire measure of current depression symptoms
Snaith-Hamilton Pleasure Scale | Administered during the baseline clinical assessment, and at the 3-month follow-up visit.
  Questionnaire 14-item scale that measures anhedonia, the inability to experience pleasure. The items cover the domains of: social interaction, food and drink, sensory experience, and interest/pastimes. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree. Either of the "disagree" responses score one point, and either of the "agree" responses score 0 points.
Perceived Stress Scale | Administered during the baseline clinical assessment, and at the 3-month follow-up visit.
  Questionnaire that measures the degree to which situations in one's life are appraised as stressful. Items were designed to assess how unpredictable, uncontrollable, and overloaded respondents find their lives to be. The scale also includes a number of direct queries about current levels of experienced stress.
State-Trait Anxiety Inventory | Administered during the baseline clinical assessment, and at the 3-month follow-up visit.
  Questionnaire that differentiates state anxiety from chronic trait anxiety symptoms.
Difficulties with Emotion Regulation Scale | Administered during the baseline clinical assessment, and at the 3-month follow-up visit.
  36-item questionnaire measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation. measures 6 empirically valid constructs related to emotion dysregulation: Non-acceptance of emotional responses, Difficulties in engaging in goal-directed behavior, Impulse control difficulties, Lack of emotional awareness, Limited access to emotion regulation strategies, and Lack of emotional clarity.
Alcohol and Drug Use Self-Efficacy Scale | Administered during the baseline clinical assessment, and at the 3-month follow-up visit.
  Questionnaire assesses self-efficacy and responses to high-risk situations that can trigger substance use.Items are grouped into negative affect, social positive withdrawal/urges, and physical/other concerns; subjects indicate how "tempted" and "confident" they would be in each situation.
Distress Tolerance Scale | Administered once during the clinical assessment.
  Questionnaire measure of emotional distress tolerance
Positive and Negative Affect Schedule-Short Form: Positive Affect | Administered once during the baseline clinical assessment.
  Questionnaire: 10-item measure of Positive Affect
Positive and Negative Affect Schedule-Short Form: Negative Affect | Administered once during the baseline clinical assessment.
  Questionnaire: 10-item measure of Negative Affect
Paced Auditory Serial Addition Task | Administered once during the baseline clinical assessment.
  mental arithmetic task with 3 trial blocks of increasing difficulty. Subjects can escape the task during block 3; latency (sec) to task termination is a primary outcome.
Brief Pain Inventory-Short Form | Administered during the baseline clinical assessment, and at the 3-month follow-up visit.
  Questionnaire measures pain severity (0=no pain; 10=pain as bad as you can imagine) and its functional impact (0=no interference; 10= interferes completely).
Current Opioid Misuse Measure | Administered during the baseline clinical assessment, and at the 3-month follow-up visit.
  Questionnaire measures risk of opioid misuse
Insomnia Severity Index | Administered during the baseline clinical assessment, and at the 3-month follow-up visit.
  Questionnaire asks about problem severity of sleep-onset, sleep-maintenance, early morning awakening, sleep satisfaction, interference with daily function, perceived impairment, and level of distress from insomnia. It has good internal consistency and concurrent validity (with polysomnography, sleep diaries, and clinician or significant-other reports), making it a valid and reliable measure of perceived sleep disturbance.
Epworth Sleepiness Scale | Administered once during the baseline clinical assessment.
  Questionnaire measures 'sleep propensity', i.e. recent likelihood of dozing or falling asleep (rather than just feeling tired) in several situations.
Psychomotor Vigilance Task | Administered once during the baseline clinical assessment.
  computerized, adaptive task (reaction time to a visual stimulus presented at random inter-trial intervals [ITI]) that will be used to assess attentional lapses; this objective, validated measure of sleepiness.
Go/No-Go Task | Administered once during the baseline clinical assessment.
  Immediate and Delayed Memory Task assesses response inhibition. Participants are told to press a button to respond to stimulus X or Y presented in an alternating pattern (Go) and to withhold responding when the pattern is broken (No-Go). We will use percentage of correctly inhibited responses for each presentation.
California Verbal Learning Test-Revised | Administered once during the baseline clinical assessment.
  Immediate and delayed memory will be assessed.
Emotional Stroop Task | Administered once during the baseline clinical assessment.
  reaction time assessment of attentional bias for both emotion-related words
Wisconsin Card Sort Test | Administered once during the baseline clinical assessment.
  number of items correct, measuring ability to shift or maintain cognitive set
Digit Symbol Substitution Test | Administered once during the baseline clinical assessment.
  Psychomotor processing speed and associative ability will be assessed.
Drug History Questionnaire | Administered once during the baseline clinical assessment.
  assesses lifetime substance use (e.g. age of initial and regular use, sequence of use of opioids and BZDs, adverse consequences of use, quit attempts.
Timeline Followback interview | Administered during the baseline clinical assessment, and at the 3-month follow-up visit
  Assesses all substance use over the past 30 days; this will generate detailed data on patterns of opioid, BZD and alcohol use (e.g. simultaneous vs. concurrent, including customized queries to determine whether using one drug primes use of another, under what affective conditions (positive, neutral, negative) substances are used together, and number of days since last use (which could influence affective, neurocognitive or behavioral measures).
Opioid /Benzodiazepine Purchasing Task | Administered once during the baseline clinical assessment.
  Hypothetical purchasing tasks (economic simulations) will assess drug demand. will be tailored to each subject's preferred opioid (e.g. heroin, oxycodone, hydrocodone) or benzodiazepine based on screening self-report.
Urinalysis | At baseline clinical assessment, and at the 3-month follow-up visit
  One urine sample will be collected and tested for opioids, methadone, cocaine, amphetamines, barbiturates, and cannabinoids using a 6-panel CLIA waived drug test. The urine sample will be collected into multi-test cups with temperature strips (CLIA Waived; temperature must be 92-96º F). Samples will be tested for opioids, methadone, cocaine, amphetamines, barbiturates (negative cutoff <300 ng/ml), and cannabinoids (negative cutoff < 50ng/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

REFERENCES:
- [Derived] Greenwald MK, Moses TEH, Lundahl LH, Roehrs TA. Anhedonia modulates benzodiazepine and opioid demand among persons in treatment for opioid use disorder. Front Psychiatry. 2023 Jan 19;14:1103739. doi: 10.3389/fpsyt.2023.1103739. eCollection 2023. PMID 36741122